CLINICAL TRIAL: NCT06503887
Title: SARS-CoV-2, Intestinal Microbiota and Mucosal Response in Lebanese Children
Brief Title: COVID-19 and Intestinal Microbiota in Children
Status: Completed | Type: Observational
Sponsor: Saint-Joseph University (Other)
Collaborators: Université Paris Cité (Other)
Responsible Party: Sponsor
Other Study IDs: CEHDF1914
Record Dates: First submitted 2024-07-11; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-04

CONDITIONS: SARS-CoV2 Infection, COVID-19, Gut Microbiota, Mucosal Response, Children
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool sample collection from enrolled children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Infected Children: collection of the stool sample within a week after a positive PCR or antigen test for SARS-CoV-2
  Interventions: Other: Stool sample collection
- recovered: represent the group of children who were infected before the stool collection
  Interventions: Other: Stool sample collection
- Controls: children enrolled and stool sample taken before the covid-19 pandemic
  Interventions: Other: Stool sample collection

INTERVENTIONS:
Other: Stool sample collection — Following the approval of the legal guardians, a stool collection container was given to the parents in order to collect the stools. Stools were kept at 4ºC for 24h max, then transported to the laboratory, aliquoted and stored at -80ºC for further analysis

SUMMARY:
SARS-CoV-2 is the causative agent of the COVID-19 pandemic. It appears to cause only mild to moderate upper respiratory symptoms in children, in addition to gastrointestinal symptoms resulting from its penetration into intestinal cells. Viral respiratory infections are often accompanied by a change in the composition of the gut microbiota (GM). Additionally, intestinal metabolites and integrity appear to be altered. This work aims to study the composition of the GM of Lebanese children, currently (n=14) and previously (n=33) infected with SARS-CoV-2 and to compare it to pre-pandemic controls (n=39). Furthermore, the correlation between the composition of the GM and the intestinal homeostasis are evaluated. Clinical data and stool samples were collected from children aged 1 month to 12 years. The bacterial profile is determined by quantitative PCR and 16S rRNA sequencing. Levels of secretory immunoglobulin A (sIgA), fecal calprotectin, beta defensin type 2 (hBD-2), short-chain fatty acids (SCFAs), tryptophan derivatives, and bile acids are also evaluated. Given the well-established relationship between the GM and the immune system, the results of this study could serve as a potential basis for the implementation of personalized nutrition and biotic supplementations aimed at restoring the host-microbiota symbiosis, pointing to the prevention and treatment of COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Within age limits
* positive PCR

Exclusion Criteria:

* metabolic disorders, hepatic disorders, immunodeficiency, allergy, autoimmune diseases, IBD, food intolerance, antibiotic administration within 3 months, pro and prebiotic administration within 3 months

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children aged between 1 month and 12 years are enrolled in the study. Sample from the control group were collected before the pandemic (for a previous study).
  For the infected and recovered children, a positive PCR test is is required for their enrollment in the study.
  All the children are healthy and do not suffer from any disease or comorbidity
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Analysis of the gut microbiota in covid-19 children | june 2024
  Quantify and analyse the composition of the gut microbiota if Lebanese infected Children

SECONDARY OUTCOMES:
Effect on covid infection on mucosal barrier | june 2024
  Evaluation of the consequences of the infection on the mucosal barrier
correlation between gut microbiota and mucosal response | september 2024
  examine the correlation between the composition of the gut microbiota and the mucosal response

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph university, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided